CLINICAL TRIAL: NCT04116840
Title: An Open-label, Sequential Parallel Group, Single Ascending Dose Following Intravenous Bolus/Infusion Administration in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MT1002 for Injection
Brief Title: Single Ascending Dose Trial to Evaluate the Safety, Tolerability, PK, and PD of MT1002 for Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MT1002-Ⅰ-C01
Record Dates: First submitted 2019-09-26; First posted 2019-10-07 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MT1002 for Injection (Experimental): Single Ascending Dose following Intravenous Bolus/Infusion Administration in Healthy Subjects
  Interventions: Drug: MT1002 for injection

INTERVENTIONS:
Drug: MT1002 for injection — Study drug will be administered by an intravenous bolus dose followed by an infusion of 4 hours.

SUMMARY:
This is an open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single dose of MT1002 for injection following intravenous bolus/infusion ascending dose administration.

DETAILED DESCRIPTION:
An initial, single dose escalation study of MT1002 for injection for injection in heathy subjects will be performed to evaluate safety, pharmacokinetics, and pharmacodynamics after intravenous bolus and infusion administration.

A total of 36 subjects (6 subjects per cohort) in 6 dose levels . At each dose level, a single sentinel subject will be dosed first. Sentinel subjects will receive a phone call at 48 hours ±4 hours to inquire about their status. If no dose-limiting toxicity is observed for 48 hours post-dose, the remaining 5 subjects in that dose level will be treated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-60 years.
2. Able and willing to give written informed consent.
3. BMI between 18.0 and 34.0 kg/m2, inclusive.
4. Subjects must be able to refrain from consuming xanthine, quinine and caffeine containing beverages, and must refrain from prolonged intensive physical exercise during the study (from 72 hours prior to dosing until the last study visit).
5. Women must be:

   * not pregnant
   * not breast-feeding
   * not planning to become pregnant during the study
6. All females must have a negative serum pregnancy test at screening and a negative urine pregnancy test at check-in on Day -1. All women must agree to use an adequate method of contraception during the study and for 30 days following the end-of-study visit.
7. Male subjects must agree to utilize a highly effective method of contraception (condom plus spermicide) during heterosexual intercourse from clinic admission until 30 days following the end of study visit.
8. Male subjects must agree to refrain from sperm donation from clinic admission until at least 30 days following the end of study visit.

Exclusion Criteria:

1. Any medical condition, clinical laboratory test or other reason which in the judgment of the Investigator or designee makes the subject unsuitable for the study.
2. Does not tolerate venepuncture or has poor venous access that would cause difficulty for collecting blood samples.
3. Has participated in an investigational drug study and received investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the screening visit or who is currently participating in another clinical trial.
4. Has experienced an acute illness within 14 days prior to the screening visit.
5. Any clinically significant abnormalities in hematology, blood chemistry and/or urinalysis lab tests at screening or at D1.
6. Known hypersensitivity to MT1002

8. History of any drug hypersensitivity that would require urgent medical care 9. Use of aspirin or any non-steroidal anti-inflammatory drug within 14 days of Day -1 10. Any serum FSH result <40mIU/mL 11. History, symptoms, or signs of cardiovascular or cerebrovascular disease. 12. History, symptoms, or signs of severe hepatic impairment. 13. HbA1c >5.7% at Screening 14. History of excessive bleeding from an injury or after surgery or dental work.

15. History of heavy or long menstrual bleeding. 16. History of blood in urine or stool or history of black stools. 17. History of easy bruising. 18. PT or aPTT > upper limit of normal at Screening or Day -1. 19. Platelet count < lower limit of normal at Screening or Day -1 20. History within the previous 3 years or current evidence of abuse of any drug, prescription or illicit, or alcohol; a positive urine screen for drugs of abuse or breathalyzer alcohol test.

21. Positive urinary test for drugs of abuse and/or alcohol breath test at Screening and/or at check-in on Day -1.

22. Supine systolic blood pressure (BP) > 130 mm Hg, diastolic BP > 80 mm Hg, respiratory rate >20 breaths per minute, pulse >90 beats per minute, or temperature >37.5º at Screening.

23. Abnormal 12-lead ECG that may jeopardize the subject's safety to participate in this study or a screening 12-lead ECG demonstrating any one of the following: heart rate (HR) > 100 beats per minute (bpm), QRS > 120 milliseconds (msec), QTcF > 450 msec, or PR > 220 msec.

24. Electrolyte abnormalities (e.g., hypokalemia or hypomagnesemia), congestive heart failure, or other medicinal products that lead to QT prolongation.

25. Any clinically significant alanine aminotransferase (ALT), alkaline phosphatase (AP), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT) or bilirubin abnormalities judged by the Investigator or designee at Screening.

27. Tobacco or nicotine users except subjects who stopped using tobacco or nicotine 90 days or more before signing the informed consent.

28. Positive Hepatitis C antibody, Hepatitis B surface antigen, or positive human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | 24 hours
  Maximum observed concentration following intravenous bolus/infusion administration of MT1002 for injection
Time to maximum concentration (Tmax) | 24 hours
  Time to maximum concentration (Tmax)
Area under the concentration-time curve (AUC) from Hour 0 to the last measurable concentration (AUC0-last) | 24 hours
  Area under the concentration-time curve (AUC) from Hour 0 to the last measurable concentration (AUC0-last)
AUC extrapolated to infinity (AUC0-∞) | 24 hours
  AUC extrapolated to infinity (AUC0-∞)
Activated clotting time (ACT) | 24 hours
  Activated clotting time (ACT)
Activated partial thromboplastin time (aPTT) | 24 hours
  Activated partial thromboplastin time (aPTT)
International normalized ratio (INR) | 24 hours
  International normalized ratio (INR)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MB, Principal Investigator — Pharmaron CPC, Inc.
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No